CLINICAL TRIAL: NCT02978443
Title: A Study to Estimate the Anti-Tumor Activity and Identify Potential Predictors of Response in Patients With Advanced Mucosal or Acral Lentiginous Melanoma Receiving Standard Nivolumab in Combination With Ipilimumab Followed by Nivolumab Monotherapy
Brief Title: A Biomarker Study in Advanced Mucosal or Acral Lentiginous Melanoma Receiving Nivolumab in Combination With Ipilimumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Georgetown University (Other)
Collaborators: Melanoma Research Foundation Breakthrough Consortium (Other); Bristol-Myers Squibb (Industry); University of Colorado, Denver (Other); University of California, San Francisco (Other); Vanderbilt University (Other); Columbia University (Other); University of Pittsburgh (Other); Yale University (Other); M.D. Anderson Cancer Center (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Memorial Sloan Kettering Cancer Center (Other); Northwestern University (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0420; CA209-763 (Other: Bristol-Myer Squibb (BMS))
Record Dates: First submitted 2016-11-23; First posted 2016-12-01 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Acral Lentiginous Melanoma; Mucosal Melanoma
Keywords: Melanoma; Mucosal; Acral Lentiginous; Ipilimumab; Nivolumab; Anti-tumor; Potential Predictors; Opdivo; Yervoy
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab-Ipilimumab Combination Therapy (Experimental): All patients will receive nivolumab administered IV over 60 minutes at 1 mg/kg combined with ipilimumab administered IV over 90 minutes at 3 mg/kg every 3 weeks for 4 treatment cycles (Induction) then continue with nivolumab administered IV over 60 minutes at 3 mg/kg every 2 weeks until progression, intolerable toxicity, or a maximum of 48 weeks, whichever comes first (Maintenance). Patients exhibiting complete response (CR) should continue nivolumab monotherapy at least 12 weeks beyond documentation of CR, if possible.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — nivolumab administered IV over 60 minutes at 1 mg/kg every 3 weeks for 4 treatment cycles (Induction) then continue with nivolumab administered IV over 60 minutes at 3 mg/kg every 2 weeks
  Other Names: BMS-936558; Opdivo
Drug: Ipilimumab — ipilimumab administered IV over 90 minutes at 3 mg/kg every 3 weeks for 4 treatment cycles (Induction)
  Other Names: BMS-734016; Yervoy

SUMMARY:
Participants with advanced or metastatic mucosal melanoma (cohort A) and acral lentiginous melanoma (cohort B) eligible for treatment with nivolumab in combination with ipilimumab followed by nivolumab therapy will submit tissue blocks from tumors of malignant melanoma for histopathology review and immunohistochemistry analysis at Georgetown University-Lombardi Comprehensive Cancer Center. Pretreatment blood will be drawn and stored in the Melanoma Research Foundation Breakthrough Consortium Virtual Repository at each participating institution. At the end of participation, samples will be sent to Georgetown University-Lombardi Comprehensive Cancer Center for processing and storage. An optional pretreatment biopsy of an accessible tumor lesion will be performed in a subset of enrolled patients. Patients will receive nivolumab in combination with ipilimumab according to the standard FDA approved treatment regimen.

DETAILED DESCRIPTION:
Immunotherapy with HD-IL-2 has produced durable benefit in 10% of patients with metastatic cutaneous melanoma. The antitumor activity of IL-2 has been limited at least in part by immunosuppressive and immune-regulatory forces within the tumor microenvironment. Antibodies against CTLA4 (e.g. ipilimumab), PD1 and its ligand (PD-L1) produced long-term benefit in approximately 20-40% of patients with advanced melanoma. In addition, the combination of ipilimumab with the anti-PD1 antibody, nivolumab, has shown tumor responses in up to 60% of patients with advanced melanoma. These findings have led to FDA approval of ipilimumab and nivolumab as an indication for treatment of patients with advanced melanoma and nivolumab for other cancers. While these data are exciting, only a few patients enrolled to the prior studies had metastatic MCM or ALM. There is no prospective immunotherapy studies conducted in MCM or ALM-specific population. Therefore the activity of the ipilimumab + nivolumab combination in these subsets or patients remains unknown

Reliable predictive biomarkers for the use of immune checkpoint inhibitors are needed to identify pretreatment those patients most likely to respond and early on in treatment assays could help identify mechanisms of tumor response and resistance necessary to improve therapy. Although tumor PD-L1 expression in tumor confers higher treatment response rate, responses to nivolumab or nivolumab + ipilimumab alone were noted in 55% and 41% of patients, respectively, with PD-L1- tumors. Therefore, more reliable predictive biomarkers are needed.

Recently, extensive studies on metastatic colorectal cancer have demonstrated that a new scoring system as well as density of immune cells infiltrates at the center of the tumor and its invasive margin, described as Immunoscore, could accurately separate a group of patients with high Immunoscore with improved DFS, and OS from those with low Immunoscore where the histopathological staging system cannot. A recent study has also demonstrated relationship between degree of pre-treatment CD8+ tumor infiltrating lymphocytes (TILs) infiltration and PD-L1 expression at the invasive margin of the advanced cutaneous melanoma and improved long-term clinical benefits in patients with advanced melanoma who received pembrolizumab monotherapy. Further, there appeared to be an association between tumor response and clonality of the immune infiltrate based on a next-generation sequencing method used to evaluate T-cell receptor rearrangement pre- and in response to checkpoint inhibitor therapy. Also, high mutational burden correlated with overall survival in patients with cutaneous melanoma treated with ipilimumab or lung cancer treated with anti-PD1. However, the biology of MCM and ALM are distinct from cutaneous melanoma at multiple levels. Consequently, the utility of predictive biomarkers developed for cutaneous melanoma remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed MCM or ALM that is metastatic or unresectable.
* Patients must be eligible to receive nivolumab in combination with ipilimumab treatment per institutional guidelines.
* Patients must have a tissue block (or 20 unstained slides) available with adequate tumor to perform multiplex immunohistochemistry and nucleic acids analyses ( i.e. whole exome sequencing) Patients with only a previous fine-needle aspirate are ineligible for enrollment.
* Patients must be willing to donate a small amount of whole blood prior to treatment and during treatment for laboratory analysis.
* Patients must give informed consent prior to initiation of therapy.
* Patients must be ambulatory with good performance status (ECOG 0 or 1)

Exclusion Criteria:

* Patients who do not have available tissue for immunohistochemistry and nucleic acids analyses.
* Patients who have received prior immunotherapy for unresectable or metastatic disease.
* Patients with untreated brain metastases, leptomeningeal disease, or seizure disorders are ineligible. Patients with a history of brain metastases must have completed treatment (i.e. surgery or radiation) 1 month prior to enrollment and have no evidence of disease or edema on brain CT or head MRI.
* Patients with inadequate tissue for analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suthee Rapisuwon, MD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - John Theurer Cacner Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab-Ipilimumab Combination Therapy
Started | 14
Completed | 0
Not Completed | 14
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 3
Not completed — Disease Progression on study | 6
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Switch to alternative therapy | 1
Not completed — Refused further treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab-Ipilimumab Combination Therapy
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) With Mucosal Melanoma (MCM)
Description: ORR, defined as complete response [CR] + partial response [PR] per RECIST 1.1 criteria and to compare this response rate to the response rate of patients with "good" molecular predictive features
Time Frame: 24 months
Population: patients with mucosal melanoma (MCM)
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab-Ipilimumab Combination Therapy
Number analyzed (Participants) | 9
Participants | 1

2. Secondary Outcome: Objective Response Rate With Acral Lentiginous Melanoma (ALM)
Description: as for outcome 1
Time Frame: 24 months
Population: patients with with acral lentiginous melanoma (ALM)
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab-Ipilimumab Combination Therapy
Number analyzed (Participants) | 4
Participants | 1

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from the date of treatment initiation until the date that disease progression criteria are met or the date death without progression, or is censored at the date of last disease assessment without evidence of progression.
Time Frame: 33 months
Measure: Median (Full Range); unit: days
Arm/Group | Nivolumab-Ipilimumab Combination Therapy
Number analyzed (Participants) | 13
days | 127 [12 to 995]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is calculated from the date of treatment initiation to the date of death, or censored at date of last contact.
Time Frame: 44 months
Measure: Median (Full Range); unit: days
Arm/Group | Nivolumab-Ipilimumab Combination Therapy
Number analyzed (Participants) | 13
days | 567 [12 to 1312]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from time of consent through 100 days of discontinuation of treatment; up to 1 year. All Cause mortality was assessed from start of treatment through up to 44 months.
Arm/Group | Nivolumab-Ipilimumab Combination Therapy
All-Cause Mortality (participants affected / at risk) | 9/13
Serious Adverse Events (participants affected / at risk) | 7/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab-Ipilimumab Combination Therapy (N=13)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) — biliary obstruction due to biliary stent migration
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — Disease Progression
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab-Ipilimumab Combination Therapy (N=13)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) — decreased cerumen/cerumen obstruction
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — dark stools
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Generalized Body aches
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Radiculopathy
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Spondylosis
Infusion related reaction (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (12)
Alkaline phosphatase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 4 (6)
Blood bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2) — Thrombocytopenia
Lymphocyte count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Hepatobiliary disorders, other- specify (Hepatobiliary disorders) | 1 (1) — Elevated LFT

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/43/NCT02978443/Prot_SAP_000.pdf